CLINICAL TRIAL: NCT01184235
Title: Actigraphic, Observational, Psychometric and Biological Measurement of Psychopharmacological Treatment Response
Brief Title: Multidimensional Measurement of Psychopharmacological Treatment Response
Status: Completed | Type: Observational
Sponsor: Child Psychopharmacology Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Act3
Record Dates: First submitted 2010-08-12; First posted 2010-08-18 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Autism Spectrum Disorders; Mood Disorders; Sleep Disorders; Attention Deficit Disorders
Keywords: Circadian Disorders; Autism Spectrum Disorders; Mood Disorders; Executive Functioning; Pediatric Mood Disorders
MeSH Terms: conditions — Autism Spectrum Disorder; Mood Disorders; Sleep Wake Disorders; Attention Deficit Disorder with Hyperactivity | interventions — Antipsychotic Agents; Antidepressive Agents; Central Nervous System Stimulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Autism Spectrum Disorders: This group will include those receiving or anticipating receiving pharmacological intervention whose primary diagnosis is Autism Spectrum Disorder
  Interventions: Drug: Pharmacological Intervention
- Attention Deficit Hyperactivity Disorder: This group will include those receiving or anticipating receiving pharmacological intervention whose primary diagnosis is Attention Deficit Hyperactivity Disorder.
  Interventions: Drug: Pharmacological Intervention
- Unaffected 1st Degree Relatives: This group will include unaffected, non treated first degree relatives of this study's subjects receiving or anticipating receiving pharmacological intervention.
- Mood Disorders: This group will include those receiving or anticipating receiving pharmacological intervention whose primary diagnosis is mood disorder.
  Interventions: Drug: Pharmacological Intervention

INTERVENTIONS:
Drug: Pharmacological Intervention — This study will include those anticipating or receiving any pharmacological intervention
  Other Names: antipsychotics; antidepressants; mood stabilizers; stimulants; NMDA antagonists
  Groups: Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorders; Mood Disorders

SUMMARY:
The study examines actigraphic, observational, psychometric and associated repeated measurements obtained prior to and during psychopharmacological treatment.

DETAILED DESCRIPTION:
Baseline actigraphic measurements, multi-symptom operationally defined observations and psychometric data will be established and repeated to measure treatment response. Additional biological and biometric measures that have potential to further characterize the cohorts under study or treatment response will be collected as practical and when possible.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of:
* Autism Spectrum Disorder
* Mood Disorder
* Attention Deficit Hyperactivity Disorder
* Unaffected First Degree Relative of Study Subject
* Anticipation of pharmacological intervention or current pharmacological intervention

Exclusion Criteria:

Inability to wear an actigraphy watch

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults, male or female receiving or anticipating pharmacological intervention and their non-affected first degree relatives will be invited to participate based on institutional actiwatch availability. Since children are the focus of the Child Psychopharmacology Institute they will be the primary recruitment focus, however, adult subjects may include non-affected first degree relatives or others who represent designated cohort groups and will be accepted based on actiwatch availabilty.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Actigraphic Measurement | Three week actigraphic measurement periods
  Actigraphic measurements are recorded every 30 seconds during three week measurement periods. The actigraphic measurements will be made utilizing an Actiwatch (AW-64 Phillips-Rispironics, Inc.), placed on the subject's non-dominant wrist. The measurements will occur every thirty seconds for approximately 21 consecutive days. Actigraphic measurements collected at this frequency reflect circadian patterns of interest; discern sleep states and characterize activity and activity patterns.

SECONDARY OUTCOMES:
Operationally Defined Observations | Randomly repeated treatment course observational measurements during actigraphic measurement periods
  The Systematic Observation Scale™ utilizes operationally defined symptoms that are presented to the primary observer (self or parent) for determination regarding the percentage of time symptoms are present. Target symptoms will be defined at baseline. Systematic Observation Scale measurements will be obtained at baseline and weekly post-treatment for periods defined as treatment initiation, treatment adjustment or treatment-course longitudinal.

CONTACTS AND LOCATIONS:
Overall Officials: Bill J Duke, M.A., Ph.D., Principal Investigator — Child Psychopharmacology Institute; Robert D Staton, Ph.D., M.D., Principal Investigator — Child Psychopharmacology Institute
Locations (1):
- Child Psychopharmacology Institute, Fargo, North Dakota, United States

REFERENCES:
- [Result] B. Duke and D. Staton,